CLINICAL TRIAL: NCT04134819
Title: Missing Microbes in Infants Born by Caesarean Section: Antenatal Antibiotics and Mode of Delivery
Brief Title: Missing Microbes in Infants Born by Cesarean Section
Acronym: MiMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: Dupont Applied Biosciences (Industry)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Consultant Neonatologist, University College Cork
Other Study IDs: APC088
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: C Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with microbial DNA not human DNA. The following samples will be collected: Faecal (adult), faecal (infant), urine (infant), saliva cortisol (adult and infant), hair (adult and infant), breast milk, vaginal swab or skin swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Vaginally Delivered Babies- No antibiotic treatment: Adult healthy pregnant females (in total 400) as well as their infants will be recruited. It is expected 67% of babies will be vaginally delivered and that 60% will not have antibiotic treatment during pregnancy. This will be up to 161 mother/infant dyads.
- Vaginally Delivered Babies- antibiotic treatment: It is expected based from previous hospital statistics that 67% of babies will be vaginally delivered and 40% of these women will be treated with antibiotics during pregnancy. This could be up to 107 mother/infant dyads.
- C-section Delivered Babies- No antibiotic treatment: It is expected based from previous hospital statistics that 33% of babies will be delivered by C section and that 60% will not have antibiotic treatment during pregnancy. This will be up to 80 mother/infant dyads All C Section women (including emergency C Section) will be treated with IV Cefazolin at the time of incision, in theatre, to prevent internal wound infection.
- C-section Delivered Babies- antibiotic treatment: It is expected based from previous hospital statistics that 33% of babies will be delivered by c section and 40% of these women will be treated with antibiotics during pregnancy. This could be up to 52 mother/infant dyads .All C Section women (including emergency C Section) will be treated with IV Cefazolin at the time of incision, in theatre, to prevent internal wound infection.

SUMMARY:
General adult healthy pregnant females in total 400, as well as their infants will be recruited. It is expected 67% will be vaginally delivered and 33% will be C Section deliveries. It is expected that of these groups that 40% of these women will be treated with antibiotics during their pregnancy. All C Section women (including emergency C Section) will be treated with IV Cefazolin at the time of incision, in theatre, to prevent internal wound infection.

Primary objective The effect of maternal antibiotic administration during pregnancy upon the development of the intestinal microbiota until the age of two years; of C-section delivered infants compared to C-section delivered infants born to non-antibiotic treated pregnant women. To develop a cohort of vaginally delivered infants to isolate the 'missing microbes' (intestinal) in the groups above.

Secondary objective

The effect of maternal antibiotics on the developing infant by:

* Anthropometric assessment: Body weight and Body length
* Bayley scale of infant development test at age 2 years

Ancillary

* To isolate and characterise bacterial strains from fresh healthy infant faeces that are altered in the stools from C-section delivered and antibiotic treated infants and compared to vaginally delivered infants.
* The effect of maternal antibiotic treatment on the human milk microbiome during lactation
* Stress hormone levels of mothers and infants
* Mental health questionnaire of mothers
* Food frequency questionnaire of mothers Exploratory
* To identify bacterial strains that can be further developed into probiotic products to help replenish depleted microbiota in the infant gut, born by C Section and or treated with antibiotics

DETAILED DESCRIPTION:
The intestinal microbiota in early life plays a major role in infant health and development, impacting on maturation of the immune system, protection against pathogens, and influencing the long-term metabolic welfare of the host. The acquisition of microbial strains from mother to infant may occur through multiple different pathways, including the birth canal (and the proximity of the birth canal to the anus), contact between mothers and infant during parental care and through breast milk. From birth through to the initial stages of weaning, microbial composition has a significant impact on the infant gut. Recent advances in culture-independent sequencing technologies has allowed for the identification of key microbial species involved in the initial colonization process, including those facultative anaerobes such as Streptococcus, Staphylococcus and Enterobacter spp. Thus, the microbiome of vaginally born, exclusively breast fed infants at term, with no previous exposure to antibiotics either directly or indirectly from the mother, could be considered the "gold standard". Breast milk, a natural prebiotic source provides the optimal active ingredients for the growth of beneficial microbial species. A disturbance in the balance of microbial inhabitants can affect human host biology in many ways. Immune, endocrine, cognitive, as well as metabolic functions can be influenced by the microbial communities present; subsequently implicating future health outcomes such as insulin resistance, allergic diseases, depression and perhaps even autism. Beneficial microbial species and its associated bioactive compounds, which may restore overall gut health are thus of interest for infant nutrition, which when administered, may help treat or prevent a microbial disturbance in the gastrointestinal environment and have long term health benefits.

The gut microbiota appears to influence the development of emotional behaviour, stress- and pain-modulation systems, and brain neurotransmitter systems. Additionally, microbiota perturbations by probiotics and antibiotics exert modulatory effects on some of these measures have been seen in adult animal models. Current evidence suggests that multiple mechanisms, including endocrine and neurocrine pathways, may be involved in gut microbiota-to-brain signalling and that the brain can in turn alter microbial composition and behaviour via the autonomic nervous system. Therefore, another aspect of the work will involve studies addressing microbe to brain signalling to identify and develop commensal probiotic consortium (mixed strains and possibly mixed strains/ingredient mixes) products underpinned by the necessary science suitable for development of probiotics targeted at the microbiota-gut-brain axis, a bidirectional communication between the gastrointestinal system and the brain, which regulates brain function and plays a crucial role in mood control. It is well established that probiotic intervention, at least in mice, can improve mood and reduce anxiety in various models of stress. Despite confounding evidence, the mood enhancing impact of probiotic intervention observed in murine studies are not always translated in humans.

Babies born by C-section get the greatest benefit from breastfeeding, and often these mothers are taking antibiotics for 1-2 weeks post-delivery. Antibiotics are administered at time of incision (for both elective and emergency sections) to prevent internal wound infection. While human milk itself could be a source of bacteria for the developing infant, thereby influencing microbial intestinal colonization following birth, many questions remain about the impact of nutrition during pregnancy and lactation, source of the 'milk microbiome' and its impact on the establishment of the infant gut microbiota. A limited number of studies have examined the microbial communities present within breast milk and tracked alterations in microbial diversity throughout the lactation period. However, in a recent study, the investigator's group reported the presence of a core breast milk microbiome using Illumina MiSeq sequencing to detect 12 dominant genera in lactating mothers (n=10), constituting 81% of the taxa present over the first 6 weeks of life. A number of frequently shared taxa, including Bifidobacterium, Lactobacillus, Staphylococcus and Enterococcus were common in both breast milk and infant faeces during the first 3 months of life, and culture-dependent analysis identified identical strains of Bifidobacterium breve and Lactobacillus plantarum present in both breast milk and infant faeces, confirming the concept of maternal-infant transmission. Similar findings have been reported using randomly amplified polymorphic DNA (RAPD) and/or multi-locus sequence typing (MLST) to identify identical genomic patterns of Bifidobacterium and Lactobacillus present in breast milk and corresponding infant faeces.

Antibiotic treatment throughout pregnancy accounts for 80% of prescribed medications during pregnancy. The Mayo Clinic describes amoxicillin, ampicillin, clindamycin, erythromycin, penicillin and nitrofurantoin as being generally considered safe during pregnancy. Tetracyclines can damage a woman's liver during pregnancy, and trimethoprim + sulfamethoxazole (commonly used together to treat UTIs) may be linked with an increased risk of birth defects. Considering that it is now accepted that optimal establishment of the gut microbiota is highly desirable for normal human development, the risk is that antibiotic usage during pregnancy may have undesirable effects on the maternal vaginal and milk microbiome, with knock-on negative impact on the early infant microbiome. It is estimated that one in five pregnant women in Europe is prescribed at least one course of antibiotics during pregnancy; in the United States, this rate is double. In the case of proven maternal infection, narrow spectrum antibiotics should be preferred due to their less extensive effects on the microbiome, taking into account the association of prenatal antibiotics with increased risk of childhood atopic disease, epilepsy, and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females of age 22 to 40 years
* Singleton pregnancy
* Infants born within the Cork University Maternity Hospital
* Women who are intending to exclusively breast feed their infant for a minimum of 6 weeks
* Mothers who give birth to full term infants greater than 35 weeks' gestation
* Infants who are born healthy with no underlying illness, syndrome or chronic disease
* Participants who agree to maintain their usual dietary habits throughout the trial period
* Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
* Consent to participate in the study and willing to comply with the protocol and study restrictions.

Exclusion Criteria:

* Sick infants who are admitted to the neonatal unit
* Stillbirth or live birth where the baby is born alive but dies shortly after.
* Infants born less than 35 (34 weeks +6 days) weeks gestation
* Infants who are formula fed exclusively before 6 weeks of age
* Mothers with insulin dependent gestational diabetes)
* Mothers and infants who will live more than 45 minutes (driving) from hospital on discharge.
* Self-declare history of alcohol abuse (for females: >3 drinks on any single day and >7 drinks per week
* Self-declare use of illicit drugs
* Participants under administrative or legal supervision.
* Participation in another study with any investigational product within 60 days of screening

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Mothers are recruited to the study based on gender Gender is not a criteria for Infants
Study Population: Pregnant women will be approached during the 3rd trimester at antenatal clinics. An arrangement will be made to meet them at their next hospital visit to obtain consent and stool sample. An information leaflet about the study will be given & the aim of the study will also be explained to them by the research nurse/researcher. They will be given time to make an informed decision & to ask questions regarding the study; if they wish to participate with their infant, the putatively eligible participants must sign the informed consent form (ICF) before beginning any study-related activities. Hereafter an inclusion/exclusion checklist will be completed. Participants will complete a food frequency questionnaire and mental health questionnaire during the screening visit as well as during visit 6.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Differences in intestinal microbiota between C-section delivered infants exposed to maternal antibiotic administration during pregnancy and non-exposed infants | 2 years
  The effect of maternal antibiotic administration during pregnancy upon the development of the intestinal microbiota until the age of two years; of C-section delivered infants compared to C-section delivered infants born to non-antibiotic treated pregnant women. To develop a cohort of vaginally delivered infants to isolate the 'missing microbes' (intestinal) in the groups above.

SECONDARY OUTCOMES:
The effect of maternal antibiotics on the developing infant by: | 24 weeks and 12 months
  Weight (kg)
The effect of maternal antibiotics on the developing infant by: | 24 weeks and 12 months
  Length cm
The effect of maternal antibiotics on the developing infant by: | 24 weeks and 12 months
  head circumference of infant. cm

OTHER OUTCOMES:
To isolate and characterise bacterial strains from fresh healthy infant faeces | birth, one week post birth, 4 weeks, 8 weeks, 24 weeks, 12 months, 18 months and 24 months.
  Stool microbiotia
The effect of maternal antibiotic treatment on the human milk microbiome during lactation | 1, 4, 8 weeks, 6 months and 12 months
  Breast milk Microbiotia
Stress hormone levels of mothers and infants | 4 weeks
  Hair cortisol levels
Edinburgh postnatal depression scale | 8 weeks
  Questionnaire based
Food frequncy questionnaire | 6 months
  Quetsionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eugenen M Dempsey, PhD MD, Principal Investigator — APC Microbiome Ireland, University College Cork, Ireland.
Locations (1):
- Cork University Maternity Hospital, APC Microbiome Ireland, University College Cork, and Teagasc Food Research Centre, Moorepark, Fermoy, Co. Cork. IRELAND, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warda AK, Dempsey EM, Forssten SD, Ryan CA, Cryan JF, Patterson E, O'Riordan MN, O'Shea CA, Keohane F, Meehan G, O'Connor O, Ross RP, Stanton C. Cross-sectional observational study protocol: missing microbes in infants born by caesarean section (MiMIC): antenatal antibiotics and mode of delivery. BMJ Open. 2022 Nov 2;12(11):e064398. doi: 10.1136/bmjopen-2022-064398. PMID 36323464